CLINICAL TRIAL: NCT03022890
Title: Pilot Study of Yoga vs. Health Education for Chronic Pain in Persons Receiving Opioid Agonist Therapy
Brief Title: Study of Yoga vs. Health Education for Chronic Pain in Persons Receiving Opioid Agonist Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Butler Hospital (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R34AT009432 (NIH); R34AT009432 (NIH)
Record Dates: First submitted 2017-01-05; First posted 2017-01-18 (Estimated); Last update posted 2019-08-09 (Actual); Status verified 2019-08

CONDITIONS: Opioid-Related Disorders; Pain, Chronic
MeSH Terms: conditions — Opioid-Related Disorders; Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hatha yoga (Experimental): 12 weeks of hatha yoga classes, once per week
  Interventions: Behavioral: hatha yoga
- Health education (Placebo Comparator): 12 weeks of health education classes, once per week
  Interventions: Behavioral: health education

INTERVENTIONS:
Behavioral: hatha yoga — 12 weeks of hour-long gentle hatha yoga classes
  Arms: Hatha yoga
Behavioral: health education — 12 weeks of hour-long classes on nutrition, sleep, coping with pain, and other health educaiton topics
  Arms: Health education

SUMMARY:
The Specific Aims of this treatment development research are:

To conduct a pilot randomized clinical trial (n = 40) of hatha yoga vs. a health education group (attention control) for persons with chronic pain who are taking methadone maintenance therapy (MMT) or bupreonorphine (BUP) for opioid use disorder maintenance treatment. Participants will be enrolled in the active intervention for 3 months, and then be followed for 6 months afterwards. Investigators' aims are:

1. To assess feasibility and acceptability of both the yoga class and the health education control group. Investigators will assess credibility of the assigned intervention and expectancy for improvement for both groups at baseline, program satisfaction following program participation, participant adherence (class attendance rate and amount of home practice corresponding to assigned study arm), and instructor fidelity to the manuals. Investigators will conduct structured interviews following program participation to understand specific aspects of both programs considered attractive, useful, or not useful; we will solicit suggestions for improvements as well.
2. To assess safety, investigators will track all adverse events in a structured fashion. Investigators do not expect to see any serious adverse events definitely or probably related to study participation.
3. To assess feasibility of research procedures, investigators have benchmarks for recruitment rate, retention for study assessments, and reliability of instructor fidelity measures.

DETAILED DESCRIPTION:
Chronic pain is a significant problem for people receiving opioid agonist therapy (OAT) for opioid dependence - i.e., buprenorphine/ naloxone (BUP) and methadone maintenance treatment (MMT). At least half of patients receiving BUP and MMT report chronic pain. In this population, chronic pain is associated with pain-related disability, psychiatric problems, physical problems, and increased likelihood of misuse of opioids or other illicit drugs, often leading providers to terminate treatment. Several issues complicate pharmacologic pain treatment in OAT patients, including opioid-induced hyperalgesia, increased tolerance of opioids, illicit drug use, use of benzodiazepines and alcohol, and patients' own fears about medications and addiction. Further, providers may have insufficient education regarding pain management in OAT patients, and have difficulty resolving the seeming inconsistencies between a pain management approach and an addiction management approach. There are few studies of non-pharmacologic treatment approaches to pain in OAT patients. Cognitive-behavioral therapy may be efficacious for treating pain across a range of chronic pain conditions, but studies of CBT for pain relief amongst substance abusers are rare.

Hatha yoga may be a beneficial adjunctive approach to treating chronic pain, decreasing pain-related disability, and preventing opioid misuse during OAT. Hatha yoga involves breath control (pranayama), physical postures (asanas), and meditation (dhyana). Yoga includes benefits of relaxation training, physical activity, and mindfulness training in a single unified practice. Further, yoga is a non-pharmacologic approach to pain, and therefore avoids many of the problems surrounding pharmacologic treatment of chronic pain in people receiving OAT. Yoga is a promising approach for treatment of chronic pain in people enrolled in OAT because: 1) yoga has evidence supporting its ability to reduce pain-related disability and pain severity in other populations; 2) there are plausible cognitive/affective and behavioral mechanisms by which yoga may reduce chronic pain, decrease pain-related disability, and reduce opioid misuse; 3) yoga is increasingly popular and available; 4) yoga can be a complement to other types of pain and substance use treatment; 5) yoga students may like the focus on improving overall health and well-being rather than on "fixing" a problem.

Thus, the investigators propose to conduct treatment development research that would prepare us to study whether yoga (vs. a health education control group) might be an efficacious adjunctive treatment for pain in people enrolled in OAT for opioid use disorders.

The specific aims are:

To conduct a pilot randomized clinical trial (n = 40) of hatha yoga vs. a health education group (attention control) for persons with chronic pain who are taking methadone maintenance therapy (MMT) or bupreonorphine (BUP) for opioid use disorder maintenance treatment. Participants will be enrolled in the active intervention for 3 months, and then be followed for 6 months afterwards. Investigators' aims are:

1. To assess feasibility and acceptability of both the yoga class and the health education control group. Investigators will assess credibility of the assigned intervention and expectancy for improvement for both groups at baseline, program satisfaction following program participation, participant adherence (class attendance rate and amount of home practice corresponding to assigned study arm), and instructor fidelity to the manuals. Investigators will conduct structured interviews following program participation to understand specific aspects of both programs considered attractive, useful, or not useful; we will solicit suggestions for improvements as well.
2. To assess safety, investigators will track all adverse events in a structured fashion. Investigators do not expect to see any serious adverse events definitely or probably related to study participation.
3. To assess feasibility of research procedures, investigators have benchmarks for recruitment rate, retention for study assessments, and reliability of instructor fidelity measures.

Investigators will use information collected from participant interviews as well as feedback from yoga and health education instructors and experts in addiction, chronic pain, and yoga to make modifications to interventions or research procedures intended to improve acceptability, feasibility, and safety whenever possible. This project will provide investigators with materials, experience, and pilot data needed for the next stage of this line of research, namely, a fully powered randomized clinical trial. Hatha yoga has a potential to decrease pain-related disability, pain severity, and opioid misuse in this population of people with difficult-to-treat chronic pain.

ELIGIBILITY:
Inclusion Criteria:

1. Enrolled in methadone maintenance treatment or buprenorphine treatment for 3 or more months;
2. Plan to continue this treatment for next 6 months;
3. Chronic pain, defined as pain duration for at least three months (Dworkin et al., 2012), a mean score of 4 or higher on the BPI Pain Interference Scale (C. S. Cleeland & Ryan, 1994), and pain severity of 4 or higher on a Visual Analog Scale (0-10) indicating "worst pain in the last week"(Breivik et al., 2008; Jensen, Chen, & Brugger, 2003);
4. No current psychosis;
5. Do not anticipate have surgery in the next 6 months;
6. Not currently taking yoga classes, not practicing yoga once per week or more often at home;
7. Not engaging in meditation once per week or more often;
8. Medically cleared by a primary care physician or SSTAR's OAT physician for mild-moderate physical activity (this is the only criterion NOT required for Phase 1 participants);
9. Not pregnant;
10. Aged 18 or older;
11. Proficiency in English sufficient to engage in informed consent in English and understand classes taught in English.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2018-11-16 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Client Satisfaction Questionnaire | 3 months
  satisfaction with interventions
Credibility Expectancy Questionnaire (CEQ) | 1 month
  credibility of interventions and expectancy of improvement due to interventions
Participant adherence | 3 months
  Class attendance
Participant homework adherence | 3 months
  Homework questionnaire
Instructor manual fidelity checklist | 3 months
Systematic Assessment of Treatment-Emergent Events - General Inquiry | 3 months
  used for documenting any adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Stanley Street Treatment and Resources, Fall River, Massachusetts, United States

REFERENCES:
- [Derived] Uebelacker LA, Van Noppen D, Tremont G, Bailey G, Abrantes A, Stein M. A pilot study assessing acceptability and feasibility of hatha yoga for chronic pain in people receiving opioid agonist therapy for opioid use disorder. J Subst Abuse Treat. 2019 Oct;105:19-27. doi: 10.1016/j.jsat.2019.07.015. Epub 2019 Jul 24. PMID 31443887